CLINICAL TRIAL: NCT02117011
Title: Effects of a Structured Exercise Program on Cancer-Related Fatigue in Women Receiving Radiation Therapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012-1377 Georgetown Lombardi
Record Dates: First submitted 2014-03-26; First posted 2014-04-17 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity (Other): An 8-week structured, moderate-intensity aerobic training exercise regimen concurrent with their radiation therapy (N=15),
  Interventions: Other: Physical Activity
- Control (No Intervention): Patients will continue with usual care, which includes radiation treatment.

INTERVENTIONS:
Other: Physical Activity — Those participants randomized to the exercise group will be required to exercise 5 days/week for 8 weeks coinciding with the radiation treatment sessions. The exercise intervention will consist of aerobic training. Participants will be required to meet and maintain a goal of 75 min/week of aerobic exercise by using portable cycle ergometers; that is; 15 min/day for 5 days/week. The cycle ergometer consists of two cycling pedals mounted to a stationary block that allows patients to exercise while sitting. The tension on the pedals can be adjusted to provide desired tension. Patients can also move the equipment so they can use it conveniently while sitting anywhere and with any chair.
  Arms: Physical activity

SUMMARY:
Radiation therapy (RT) is often used to treat breast cancer. RT combined with breast surgery is associated with better outcomes in early stage breast cancer compared to surgery alone. Fatigue is one of the most important side effects of RT because it can decrease patients' quality of life.

Studies found that physical activity (PA) may help to improve quality of life in cancer survivors. PA has been reported to lower fatigue, anxiety, and depression. Physical inactivity over a long period of time may lead to rapid energy and physical function loss.

PA intervention studies in patients undergoing RT have included mostly White patients. There is no evidence on African American patients undergoing RT. The purpose of this study is to examine the efficacy of a structured, moderate-intensity, aerobic exercise program in reducing cancer-related fatigue in African Americans undergoing RT for localized breast cancer.

DETAILED DESCRIPTION:
* Purpose of project (one or two sentences): The objective of this study is to examine the efficacy of a structured, moderate-intensity aerobic exercise program in reducing cancer-related fatigue in African Americans undergoing RT for localized breast cancer.

2. * Study design (for example, hypothesis, research questions, standard and experimental procedures/drugs/devices or equipment, etc.):

This is a randomized clinical trial to determine the efficacy of a structured, moderate-intensity aerobic exercise program in reducing cancer-related fatigue. The study occurs at a single-center setting. There are 30 breast cancer patient/subjects in all, a portion of whom (n=15) will undergo a structured, moderate-intensity aerobic exercise delivered via a stationary cycling device (peddlers).

The study duration would be 12 months, and the administration of the study would be 8 weeks. The exercise program will be carried out at Washington Hospital Center while they wait for radiation therapy treatments.

3. * Rationale and justification for study (i.e. historical background, investigator's personal experience, pertinent medical literature, etc.): Given the widespread use of RT for treatment of early stage breast cancers, and the identification of fatigue as an important side-effect of RT, it is important to test interventions that can reduce fatigue and improve the health-related quality of life (HRQOL) among survivors. PA interventions have been shown to improve quality of life and reduce fatigue in cancer patients undergoing RT. However, most studies on PA in RT-related fatigue and HRQOL have been conducted among Whites and evidence on the efficacy of PA interventions in African Americans is lacking. Additionally, the timing of introduction of PA with respect to the RT timeline is also unclear. Finally, although preliminary studies suggest that fatigue might be related to inflammation, it is not clear whether the effect of PA on fatigue is associated with changes in inflammatory biomarkers. The purpose of this study is to test the efficacy of a structured PA intervention in reducing cancer-related fatigue among African American patients undergoing RT for breast cancer.

This study is also designed to provide pilot data on i) the acceptability of, and adherence with PA interventions in African Americans with breast cancer, and ii) the correlation of inflammation markers with fatigue and PA.

4. * Primary objective: The purpose of this study is to test the efficacy of a structured PA intervention in reducing cancer-related fatigue among African American patients undergoing RT for breast cancer.

5. * Secondary objectives: To determine the efficacy of a structured, moderate-intensity aerobic exercise program in improving HRQOL of African American patients undergoing RT for localized breast cancer.

To determine the acceptability of, and adherence with a structured, exercise intervention among African-American patients undergoing RT for localized breast cancer.

8.* Treatment Plan: 4.1 Randomization All participants (N=30) scheduled for radiotherapy will be randomized to one of the two following groups: i) a 8-week structured, moderate-intensity aerobic training exercise regimen concurrent with their radiation therapy (N=15), or ii) usual care control group (N=15). Participants will be randomized into the study by a bio-statistician once eligibility has been determined. All participants in the study will undergo radiation therapy as scheduled by their physicians. The exercise intervention will not interfere with either the dose or the timeline of their radiation therapy.

4.2 PA intervention Those participants randomized to the exercise group will be required to exercise 5 days/week for 8 weeks coinciding with the radiation treatment sessions. The exercise intervention will consist of aerobic training. Participants will be required to meet and maintain a goal of 75 min/week of aerobic exercise by using portable cycle ergometers; that is; 15 min/day for 5 days/week. The cycle ergometer consists of two cycling pedals mounted to a stationary block that allows patients to exercise while sitting. The tension on the pedals can be adjusted to provide desired tension. Patients can also move the equipment so they can use it conveniently while sitting anywhere and with any chair.

9.* Primary Study Endpoint: The primary endpoints of the study are fatigue, HRQOL, and biomarkers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* -over 18 years old or less than 75 years old.
* histologically confirmed carcinoma of the breast
* radiation therapy naive
* sedentary, as defined as <60 minutes of recreation or work requiring modest PA/week based on the 7 day physical activity recall questionnaire
* ambulatory
* negative serum pregnancy test and not planning to be pregnant in the next 3 months
* ability to understand and the willingness to sign a written informed consent.
* have breast cancer stage 0-IIIA
* completed neo-adjuvant or adjuvant chemotherapy may be concurrently receiving endocrine or HER2 directed therapy

Exclusion Criteria:

* age less than 18 years old or more than 75 years
* no histological confirmation of breast cancer
* prior breast, chest or pelvic radiotherapy
* concurrent chemotherapy
* distant metastases
* physical limitations (e.g., orthopedic, central nervous system) that contraindicate participation in a low to moderate intensity home-based walking program
* a positive pregnancy test, currently pregnant or planning to become pregnant in the next three months
* identified as the active or maintenance stage of exercise behavior
* psychiatric disorder which would render the subject unable to provide informed consent.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduce cancer-related fatigue | 8 weeks
  Fatigue Cancer-related fatigue will be determined using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) survey instrument. The FACIT-Fatigue is a 13-item subscale developed to identify a finite set of concerns specific to fatigue. The responses to the 13 items on the FACIT fatigue questionnaire are each measured on a 4-point Likert scale. Thus, the total score ranges from 0 to 52. The FACIT-Fatigue scale has been validated in patients with cancer and showed excellent internal consistency and reliability.

SECONDARY OUTCOMES:
Increase quality of life | 8 weeks
  HRQOL Cancer related HRQOL among participants in the study will be measured using the Functional Assessment of Cancer Therapy (FACT) system questionnaires.
  The Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire is one of the most widely used HRQOL instruments. It measures HRQOL in four different domains (Physical well-being, Functional well-being, Emotional well-being and Social/Family well-being). To this core questionnaire, we will add specific modules specific for breast (FACT-B) cancer. Thus, the FACT B questionnaire contains an additional series of questions specific to FACT-B some specific questions about breast cancer (37). The FACT system has a number of advantages as a method of measuring HRQOL. The questionnaires have been developed to reflect patients' concerns; moreover they are reliable, reproducible and have been validated in numerous studies. Higher scores on the FACT questionnaires reflect higher QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Lucile Adams-Campbell, Principal Investigator — Georgetown University; Pamela Randolph-Jackson, Study Director — Medstar Health Research Institute
Locations (1):
- Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia, United States